CLINICAL TRIAL: NCT02612974
Title: Randomized Controlled Clinical Evaluation of Leech Therapy in the Treatment of Knee Osteoarthritis
Brief Title: Clinical Evaluation of Leech Therapy in the Treatment of Knee Osteoarthritis
Acronym: Leech Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hamdard University (Other)
Responsible Party: Principal Investigator, M. S. M. Shiffa, Dr., Hamdard University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009/AD/JH/058
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Knee Osteoarthritis
Keywords: Qurse mafasil; leech therapy; Hirudinaria granulosa
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Leeching; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Hirudinaria granulosa and Qurse mafasil are given
  Interventions: Biological: Hirudinaria granulosa, qurse mafasil
- Group B (Active Comparator): Qurse mafasil only given
  Interventions: Biological: Hirudinaria granulosa, qurse mafasil

INTERVENTIONS:
Biological: Hirudinaria granulosa, qurse mafasil — compare the efficacy of both groups
  Other Names: leech and drug

SUMMARY:
This study has been designed to conduct as Randomized comparative clinical study.

DETAILED DESCRIPTION:
Two groups, group B received Qurse Mafasil tablet orally two tablets two times daily for 8 weeks while group A received Leech therapy once weekly for 8 weeks along with Qurse mafasil.

ELIGIBILITY:
Inclusion Criteria:

* knee osteoarthritis

Exclusion Criteria:

* pregnancy,
* lactation,
* anaemia

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
KOOS Score | end of 6 weeks
VAS | end of 6 weeks
Active Range of Motion | end of 6 weeks
Knee circumference | end of 6 weeks
15 m walking time test | end of 6 weeks

SECONDARY OUTCOMES:
KOOS subscores | end of 6 weeks